CLINICAL TRIAL: NCT06918353
Title: Construction and Evaluation of the Severity Assessment Model for AECOPD With Combination of Disease and Syndrome Based on Machine Learning
Brief Title: The Severity Assessment Model for AECOPD With Combination of Disease and Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Collaborators: The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); Henan Provincial People's Hospital (Other); Third Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); Jiangsu province hospital of TCM (Unknown); Qingdao Traditional Chinese Medicine Hospital(Qingdao Hiser Hospital) (Unknown); Xiangyang Traditional Chinese Medicine Hospital (Unknown); Yanshi People's Hospital of Luoyang City (Unknown); Shangcai County Traditional Chinese Medicine Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: Model for AECOPD
Record Dates: First submitted 2025-01-27; First posted 2025-04-09 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Keywords: Acute Exacerbation of Chronic Obstructive Pulmonary Disease; Severity Assessment Model; Combination of Disease and Syndrome; Classification and Regression Trees; Artificial Neural Network
MeSH Terms: conditions — Syndrome | interventions — Diagnosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AECOPD Patients
  Interventions: Diagnostic Test: Diagnosis and Severity Grading of AECOPD Disease

INTERVENTIONS:
Diagnostic Test: Diagnosis and Severity Grading of AECOPD Disease — Diagnosis and severity grading of AECOPD disease, as well as assessment of traditional Chinese medicine syndromes

SUMMARY:
The establishment of the AECOPD severity assessment model can quickly and accurately evaluate the condition, which is of great significance for standardizing diagnosis and treatment, improving efficacy, and improving prognosis. At the same time, it can provide ideas and methods for the research of disease assessment models in related fields.

DETAILED DESCRIPTION:
Accurate assessment of the condition is the prerequisite and basis for standardized clinical treatment. Traditional Chinese medicine has shown good efficacy and advantages in treating AECOPD, but currently there is no ideal standard for judging the severity, nor is there an accurate, practical, and TCM specific disease assessment tool. Therefore, this project integrates multidimensional variables of traditional Chinese and Western medicine, and intends to conduct research on the construction of a disease syndrome combined AECOPD disease assessment model through literature review, expert consultation, clinical investigation, and machine learning algorithms, and establish preliminary grading standards for the severity of AECOPD disease. Ultimately, it provides ideas and methods for the rapid and accurate assessment of AECOPD, standardized diagnosis and treatment, improved efficacy, improved prognosis, and research on disease assessment models in related fields.

ELIGIBILITY:
Inclusion Criteria:

* Meets AECOPD diagnostic criteria.
* Voluntarily participate in the research and sign the consent form

Exclusion Criteria:

* Individuals with severe mental disorders and cognitive impairments who are unable to communicate normally

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Investigation Questionnaire on Influencing Factors of the Severity of AECOPD | 24 hours
  The influencing factors of the severity of AECOPD were evaluated through clinical investigation questionnaires.
  Questionnaire Title: Clinical Investigation Questionnaire on Influencing Factors of AECOPD Severity.
  The questionnaire adopts the scoring method, which is divided into "very unimportant", "not important", "average", "important" and "very important", and the corresponding values are assigned as 1, 2, 3, 4 and 5 respectively.The higher the score is, the more significant the result is.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan, China